CLINICAL TRIAL: NCT04631081
Title: Occlusive Dressing vs Palmar Pedicular Island Flap in Fingertip Amputation: A Randomized Controlled Trial
Brief Title: Occlusive Dressing vs Palmar Pedicular Island Flap in Fingertip Amputation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de la main - CHUV (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-01356
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Finger Injuries
MeSH Terms: conditions — Finger Injuries | interventions — Occlusive Dressings

STUDY DESIGN:
Intervention Model Description: open-label, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occlusive dressing group (Active Comparator): patients will be evaluated on admission and benefit from wound irrigation, debridement and placement of a simple dressing with Adaptic or Jelonet, either in the Emergency department or in the Hand Surgery department. At 48 hours, they will be addressed to the Hand Surgery department to place a self-adhesive polyurethane film according. Follow-up will include a visit at 1 week for dressing change, and then weekly for further dressing change until healing
  Interventions: Other: occlusive dressing
- Surgical group (Active Comparator): In surgical group, coverage with a bipedicled palmar island flap will be performed ambulatory, either on admission if patients are directly oriented to the Hand Surgery department, or within 48h of initial visit for patients addressed from the Emergency department. The flap group will be evaluated on admission, at 48h, and 6 weeks.
  Interventions: Procedure: coverage of the fingertips with bipedicled palmar island flap

INTERVENTIONS:
Procedure: coverage of the fingertips with bipedicled palmar island flap — The initial step is wound debridement. To design the flap, a longitudinal line is drawn at the junction of the volar and dorsal parts of the finger, starting from the distal part of the proximal interphalangeal joint flexion crease. It will be harvested from distal to proximal dissecting the digital canal plane. By releasing the Cleland and Grayson ligaments, the neurovascular bundle will be dissected. On the intermediate phalange, the dorsal branch of the neurovascular bundle must be preserved to maintain blood flow to the dorsal skin. Dissection is completed at the junction between the palmo-dorsal arteries and the collateral neurovascular bundles on both sides of the finger. A triangle may be resected at the distal edge of the flap to reshape of the pulp. Bone may be resected if needed to allow tension-free closure of the distal part of the flap. No Immobilization will be necessary.
  Arms: Surgical group
Other: occlusive dressing — patients will be evaluated on admission and benefit from wound irrigation, debridement and placement of a simple dressing with Adaptic or Jelonet, either in the Emergency department or in the Hand Surgery department. At 48 hours, they will be addressed to the Hand Surgery department to place a self-adhesive polyurethane film. Follow-up will include a visit at 1 week for dressing change, and then weekly for further dressing change until healing. Skin proximal to the injury will be degreased to increase adherence of the dressing. Distally, the film leaves a pocket to collect wound exudate. During treatment, the foul-smelling liquid produced by the wound and clots collected in the occlusive dressing will not be removed. A gauze covers the occlusive dressing to protect the liquid pocket and cover potential smell.
  Arms: Occlusive dressing group

SUMMARY:
Our study aims to prospectively compare outcomes of conservative treatment (occlusive dressing) to surgery with a palmar bipedicled island flap (modified Tranquilli-Leali flap) in the management of Allen zones II-III-IV fingertip injuries in long fingers. Based on these results, the investigators intend to help provide guidelines to optimize the management, and eventually the satisfaction of these patients.

DETAILED DESCRIPTION:
The investigators intend to conduct a prospective tricentric (Hand Surgery Service in CHUV( Centre Hospitalier Universitaire Vaudois, Lausanne/ Hand Surgery Service in HUG (Hôpitaux Universitaire de Genève and Hand Surgery Service in Valais hospital, Sierre), open-label, randomized controlled trial: Occlusive dressing versus surgery in fingertips amputation.

The investigators will collect demographic data and informations about the injury including age, sex, medical history and daily medications, occupation, dominant hand, active smoking, mechanism of injury, associated injuries, time from injury to management, size and geometry (volar/transverse/dorsal) of defect, level of amputation (Allen classification), injury and repair of the nail bed.

Patients will be randomized into the occlusive dressing group or the surgical group on their first visit to the Hand Surgery department.

Both groups will have 6 months and 1-year follow-up appointment, including Ultrasound evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Allen zones II-III-IV long finger amputation.
* Trauma < 48h.

Exclusion Criteria:

* Patients who are not able to give consent
* Injuries involving the DIP joint, extensor apparatus or requiring osteosynthesis.
* Chronic dermatological disorders of the hand, immunosuppressive drugs or chemotherapy. - Patient without a consent form would be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient's satisfaction assessment according to the therapeutic option (occlusive dressing vs flap). | Enrollment in the study for one year
  Patients will be instructed to rate their satisfaction (according to different criteria: overall hand function, activities of daily living, work performance, pain, and cosmetic) by checking on a horizontal line their degree of satisfaction. After evaluation, their measurement was considered as a continuous measure (0-100 mm). Higher scores indicate better satisfaction.

SECONDARY OUTCOMES:
Objective evaluation of fingertips | Enrollment in the study for one year
  Distal fingertip sensibility (Semmens-Weinstein and 2 points discrimination test).
  Finger range of motion of the PIP(Proximal InterPhalangeal) and DIP (Distal InterPhalangeal) joints (goniometer) Coloration and pigmentation of the pulp (Dermacatch). Dexterity (Nine hole peg test). Cold intolerance using the Cold Intolerance Symptom Severity (CISS) (40). Hook nail deformity. Distal phalanx bone length before and after treatment (X-Ray). Echography multiparameters analysis: thickness of the pulp (B-mode), vascularization of the pulp (Echo-doppler), Elasticity of the pulp (Shear wave elastography) (25).
  Complications: infection rate, wound dehiscence rate, flap failure rate. Time of complete healing, time before returning to work.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Durand, MD,PhD, Principal Investigator — Service de chirurgie plastique et de la main - CHUV
Locations (2):
- Switzerland (2):
  - Hôpital du Valais, Sierre, Valais
  - HUG, Geneva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sindhu K, DeFroda SF, Harris AP, Gil JA. Management of partial fingertip amputation in adults: Operative and non operative treatment. Injury. 2017 Dec;48(12):2643-2649. doi: 10.1016/j.injury.2017.10.042. Epub 2017 Oct 31. PMID 29100662
- [Result] Conn JM, Annest JL, Ryan GW, Budnitz DS. Non-work-related finger amputations in the United States, 2001-2002. Ann Emerg Med. 2005 Jun;45(6):630-5. doi: 10.1016/j.annemergmed.2004.10.012. PMID 15940097
- [Result] van den Berg WB, Vergeer RA, van der Sluis CK, Ten Duis HJ, Werker PM. Comparison of three types of treatment modalities on the outcome of fingertip injuries. J Trauma Acute Care Surg. 2012 Jun;72(6):1681-7. doi: 10.1097/TA.0b013e318248bc8c. PMID 22695441
- [Result] Hattori Y, Doi K, Ikeda K, Estrella EP. A retrospective study of functional outcomes after successful replantation versus amputation closure for single fingertip amputations. J Hand Surg Am. 2006 May-Jun;31(5):811-8. doi: 10.1016/j.jhsa.2006.02.020. PMID 16713848
- [Result] Sebastin SJ, Chung KC. A systematic review of the outcomes of replantation of distal digital amputation. Plast Reconstr Surg. 2011 Sep;128(3):723-737. doi: 10.1097/PRS.0b013e318221dc83. PMID 21572379
- [Result] Soucacos PN. Indications and selection for digital amputation and replantation. J Hand Surg Br. 2001 Dec;26(6):572-81. doi: 10.1054/jhsb.2001.0595. PMID 11884116
- [Result] Allen MJ. Conservative management of finger tip injuries in adults. Hand. 1980 Oct;12(3):257-65. doi: 10.1016/s0072-968x(80)80049-0. PMID 7002744
- [Result] Lee LP, Lau PY, Chan CW. A simple and efficient treatment for fingertip injuries. J Hand Surg Br. 1995 Feb;20(1):63-71. doi: 10.1016/s0266-7681(05)80019-1. PMID 7759939
- [Result] Lee DH, Mignemi ME, Crosby SN. Fingertip injuries: an update on management. J Am Acad Orthop Surg. 2013 Dec;21(12):756-66. doi: 10.5435/JAAOS-21-12-756. PMID 24292932
- [Result] Ma GF, Cheng JC, Chan KT, Chan KM, Leung PC. Finger tip injuries--a prospective study on seven methods of treatment on 200 cases. Ann Acad Med Singap. 1982 Apr;11(2):207-13. PMID 6753711
- [Result] Peterson SL, Peterson EL, Wheatley MJ. Management of fingertip amputations. J Hand Surg Am. 2014 Oct;39(10):2093-101. doi: 10.1016/j.jhsa.2014.04.025. PMID 25257490
- [Result] Russell RC, Casas LA. Management of fingertip injuries. Clin Plast Surg. 1989 Jul;16(3):405-25. PMID 2673624
- [Result] Tos P, Titolo P, Chirila NL, Catalano F, Artiaco S. Surgical treatment of acute fingernail injuries. J Orthop Traumatol. 2012 Jun;13(2):57-62. doi: 10.1007/s10195-011-0161-z. Epub 2011 Oct 8. PMID 21984203
- [Result] Tang JB, Elliot D, Adani R, Saint-Cyr M, Stang F. Repair and reconstruction of thumb and finger tip injuries: a global view. Clin Plast Surg. 2014 Jul;41(3):325-59. doi: 10.1016/j.cps.2014.04.004. PMID 24996458
- [Result] de Alwis W. Fingertip injuries. Emerg Med Australas. 2006 Jun;18(3):229-37. doi: 10.1111/j.1742-6723.2006.00851.x. PMID 16712532
- [Result] Stevenson TR. Fingertip and nailbed injuries. Orthop Clin North Am. 1992 Jan;23(1):149-59. PMID 1729663
- [Result] Krauss EM, Lalonde DH. Secondary healing of fingertip amputations: a review. Hand (N Y). 2014 Sep;9(3):282-8. doi: 10.1007/s11552-014-9663-5. PMID 25191157
- [Result] Weichman KE, Wilson SC, Samra F, Reavey P, Sharma S, Haddock NT. Treatment and outcomes of fingertip injuries at a large metropolitan public hospital. Plast Reconstr Surg. 2013 Jan;131(1):107-112. doi: 10.1097/PRS.0b013e3182729ec2. PMID 22965236
- [Result] Panattoni JB, De Ona IR, Ahmed MM. Reconstruction of fingertip injuries: surgical tips and avoiding complications. J Hand Surg Am. 2015 May;40(5):1016-24. doi: 10.1016/j.jhsa.2015.02.010. Epub 2015 Mar 29. PMID 25823622
- [Result] Germann G, Rudolf KD, Levin SL, Hrabowski M. Fingertip and Thumb Tip Wounds: Changing Algorithms for Sensation, Aesthetics, and Function. J Hand Surg Am. 2017 Apr;42(4):274-284. doi: 10.1016/j.jhsa.2017.01.022. PMID 28372640
- [Result] Saraf S, Tiwari V. Fingertip injuries. Indian J Orthop. 2007 Apr;41(2):163-8. doi: 10.4103/0019-5413.32051. PMID 21139772
- [Result] Lemmon JA, Janis JE, Rohrich RJ. Soft-tissue injuries of the fingertip: methods of evaluation and treatment. An algorithmic approach. Plast Reconstr Surg. 2008 Sep;122(3):105e-117e. doi: 10.1097/PRS.0b013e3181823be0. PMID 18766028
- [Result] Hoigne D, Hug U, Schurch M, Meoli M, von Wartburg U. Semi-occlusive dressing for the treatment of fingertip amputations with exposed bone: quantity and quality of soft-tissue regeneration. J Hand Surg Eur Vol. 2014 Jun;39(5):505-9. doi: 10.1177/1753193413489639. Epub 2013 May 21. PMID 23695151
- [Result] Dumontier C, Gilbert A, Tubiana R. Hook-nail deformity. Surgical treatment with a homodigital advancement flap. J Hand Surg Br. 1995 Dec;20(6):830-5. doi: 10.1016/s0266-7681(95)80057-3. PMID 8770751
- [Result] Jafari P, Muller C, Grognuz A, Applegate LA, Raffoul W, di Summa PG, Durand S. First Insights into Human Fingertip Regeneration by Echo-Doppler Imaging and Wound Microenvironment Assessment. Int J Mol Sci. 2017 May 13;18(5):1054. doi: 10.3390/ijms18051054. PMID 28505080
- [Result] Wang L, Yuan SY. A simple and direct procedure for excision of peripheral skin above the nail root to enable nail lengthening after fingertip amputation. J Plast Reconstr Aesthet Surg. 2012 Sep;65(9):e265-6. doi: 10.1016/j.bjps.2012.03.022. Epub 2012 Apr 3. No abstract available. PMID 22475687
- [Result] Serane-Fresnel J, Lafosse T, Amsallem L, Chaves C, Delpit X, Chassat R, Masmejean EH. Fingertip reconstruction by palmar bipedicular island flap in long fingers (modified neurovascular Tranquilli-Leali flap): A dual-center study. Hand Surg Rehabil. 2020 Feb;39(1):59-64. doi: 10.1016/j.hansur.2019.11.003. Epub 2019 Nov 15. PMID 31740268
- [Result] Clark DP, Scott RN, Anderson IW. Hand problems in an accident and emergency department. J Hand Surg Br. 1985 Oct;10(3):297-9. doi: 10.1016/s0266-7681(85)80047-4. PMID 4078454
- [Result] Quell M, Neubauer T, Wagner M. [Treatment of fingertip defect injuries with a semi-occlusive dressing]. Handchir Mikrochir Plast Chir. 1998 Jan;30(1):24-9. German. PMID 9541835
- Available data/document: Individual Participant Data Set — https://www.project-redcap.org/